CLINICAL TRIAL: NCT01438112
Title: An Integrated Phase II/III, Open Label, Randomized and Controlled Study of the Safety and Efficacy of CG0070 Adenovirus Vector Expressing GM-CSF in Patients With NMIBC With Carcinoma In Situ Disease Who Have Failed BCG
Brief Title: Efficacy Study of Recombinant Adenovirus for Non Muscle Invasive Bladder Cancer
Acronym: BOND
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change in study design
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12154
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Transitional Cell Carcinoma; Bladder Cancer; Carcinoma in Situ; Carcinoma in Situ Concurrent With Papillary Tumors
Keywords: cancer; bladder cancer; transitional cell; virus; oncolytic; GM-CSF; adenovirus; intravesical; neoadjuvant; cystectomy; gene therapy; oncolytic virus; carcinoma in situ; carcinoma in situ concurrent with papillary tumors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Carcinoma in Situ; Neoplasms; Virus Diseases; Adenoviridae Infections | interventions — Oncolytic Virotherapy; Mitomycin; Interferons; valrubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CG0070 oncolytic virus (Experimental): Interventions: CG0070 oncolytic virus intravesical instillations weekly X6 with each instillation lasting 45 minutes after prior transduction agent of DDM intravesically for 15 minutes
  Interventions: Biological: CG0070 Adenovirus Vector
- Chemotherapy or Interferon (Active Comparator): Quadruple Choice as interventions
  1. Mitomycin C
  2. Interferon
  3. Valrubicin
  4. Gemcitabine
  Interventions: Other: Control Arm: Quadruple Choice

INTERVENTIONS:
Biological: CG0070 Adenovirus Vector — CG0070 adenoviral vector with GM-CSF expression given intravesically 1x10e12 viral particles for each instillations, weekly times six
  Other Names: oncolytic virus; CG0070; GM-CSF expression; adenoviral vector
  Arms: CG0070 oncolytic virus
Other: Control Arm: Quadruple Choice — Quadruple Choice Treatment Options: (same as listed above)
  Other Names: Mitomycin C; Interferon; Valrubicin; Gemcitabine
  Arms: Chemotherapy or Interferon

SUMMARY:
The use of a designed viral vector that can destroy cancer cells while leaving normal cells largely unharmed. The virus also stimulates an immunological response by producing a special factor (GM-CSF) to attract and promote the development of dendritic and T effector cells. It forms the hypothesis that this regimen may be used for people who have failed current forms of treatment and are recommended for cystectomy. It is with hope that this novel therapy will be able to delay or potentially avoid cystectomy for this patient population. Bladder instillation of this agent causes little long lasting side effects and may drastically improve the stimulation of the immune system for local cancer cell death as well as destroying those tumor cells that may have travelled to regional lymph nodes or distant organs.

DETAILED DESCRIPTION:
After the phase I/II CG0070 trial review, it became apparent that the use of CG0070 oncolytic vaccine as an intravesical agent for oncolytic lysis of tumor cells, together with the transcription of GM-CSF on site, may have distinct advantages. This first study showed excellent tumor response rates of 48-77% depending on the dose schedule administered. All of these patients had residual non-muscle invasive bladder cancer who have previously failed BCG therapy at the time of treatment.

With the addition of a transduction agent such as DDM, the intravesical instillation of CG0070 enabled uniform distribution of viral particles and exposure to the tumor during those 30-60 minutes instillations as contrast to the intra-tumor injection, intra-arterial or intravenous injection of viral particles in other oncolytic viral trials. Some or most of these delivering methodologies have obvious intrinsic imperfections and potential toxicity. This unique opportunity of an relatively easy intravesical tumor exposure is difficult to duplicate in other solid tumor models.

The replication of CG0070 in the majority of patients during the first phase I/II trial indicated tumor lysis with release of tumor specific or tumor associated antigens that have been stably expressed, in abundant quantities during tumor cell death. Release of tumor antigens have been the key elements, together with sufficient on-site GM-CSF, in stimulating strong cross-presentation and confirmation signals to the antigen presenting cells such as dendritic cells interacting with CD4+ and CD8+ T cells. This concept of a "real time" vaccine like regimen is expected to compare favorably with other forms of cancer immunotherapy treatment such as BCG in this patient population.

It is with this thought that CG0070 may find a success in this setting because of a reasonably and proven complete response rate in residual and failed BCG bladder cancer patients in the first phase I/II study (some cases with only one instillation). Of importance as well, is the demonstration in the study data of a strong GM-CSF expression during its replication phase. Those patients with carcinoma in situ disease and those with RB pathway dysfunction were particularly responsive.

It is therefore, desirable to formulate a protocol to encompass the specialty of this oncolytic vaccine and the unique intravesical delivery to prove the efficacy by a randomized controlled study. This opportunity allows a study on the CG0070's beneficial effects, if any, on the standard of care for carcinoma in situ non muscle invasive bladder cancer patients after they failed BCG therapy. The prognosis of this group presently depends mainly on early radical cystectomy, which carries a high morbidity and decrease of quality of life generally viewed as unacceptable for this group of older patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be considered high risk, with pathologically confirmed high grade disease (HG) WHO 2004
2. Patients must have pathologically-proven unresectable, primary, secondary or concurrent carcinoma in situ disease, defined by having either Ta and/or T1 with CIS, or CIS
3. Patients must have no evidence of muscle invasive disease
4. Patient need to sign a specific informed consent acknowledging that a delay of cystectomy may lead to an increase chance of progression and/or metastasis with serious or sometimes fatal consequences.
5. Patients must have received at least two or more prior courses of intravesical therapy. BCG must have been one of the prior therapies administered. Patients can have either failed BCG induction therapy within a six month period or have been successfully treated with BCG, but subsequently found to have recurrence. The standard course of intravesical therapy must include six weekly treatments (allowable range of instillations per course is 4-9). The second course of BCG can consist of three weekly treatments
6. 18 years of age or older
7. Residual disease at accrual
8. Pathologically diagnosed transitional cell (urothelial) bladder cancer (further details in 10.) patients where radical cystectomy with curative intent is indicated for superficial bladder cancer that is resistant to treatment.
9. Patients must be able to enter into the study within five weeks of their most recent diagnostic procedure, which is usually a diagnostic biopsy, a transurethral resection of bladder tumor (TURBT) procedure or other diagnostic scanning such as CT and PET procedures.
10. Histopathologically confirmed, transitional cell (urothelial) carcinoma. Urothelial tumors with mixed histology (but with <50% variant) are eligible.
11. No evidence of urethral or renal pelvis TCC by upper tract radiological imaging (e.g., intravenous pyelogram, CT urogram, or retrograde pyelogram) within the past 2 years.
12. Eastern Cooperative Oncology Group (ECOG) performance status <2.
13. Not pregnant or lactating
14. Patients with child bearing potential must agree to use adequate contraception
15. Agree to study specific informed consent and HIPAA authorization for release of personal health information
16. Adequate baseline CBC, renal and hepatic function. Renal parameters as detailed above. Absolute lymphocyte count ≥ 1,000/μL before all doses of CG0070
17. Patient to provide a tumor specimen for determination of RB pathway status

Exclusion Criteria:

1. Previous systemic chemotherapy or radiation for bladder cancer. Note: Prior immunotherapy or intravesical (administered within the bladder) chemotherapy for superficial disease is acceptable
2. No bladder cancer residual disease, such as patients that are rendered disease free by TURBT
3. History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, hypersensitivity to GM-CSF or yeast derived products, clinically meaningful allergic reactions or any known hypersensitivity or prior reaction to any of the formulation excipients in the study drugs.
4. Known infection with HIV, HBV or HCV.
5. Anticipated use of chemotherapy, radiotherapy, or other immunotherapy not specified in the study protocol while on study
6. Any underlying medical condition that, in the Investigator's opinion, will make the administration of study vaccine hazardous to the patient, would obscure the interpretation of adverse events, or surgical resection. Anticipated use of chemotherapy, radiotherapy, or other immunotherapy not specified in the study protocol while on study
7. Systemic treatment on any investigational clinical trial within 28 days prior to registration.
8. Concurrent treatment with immunosuppressive or immunomodulatory agents, including any systemic steroid (exception: inhaled or topically applied steroids, and acute and chronic standard dose NSAIDs, are permitted). Use of a short course (i.e., ≤ 1 day) of a glucocorticoid is acceptable to prevent a reaction to the IV contrast used for CT scans.
9. Immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry.
10. History of prior experimental cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine)
11. History of partial cystectomy in the setting of bladder cancer primary tumor.
12. History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, hypersensitivity to GM-CSF or yeast derived products, clinically meaningful allergic reactions or any known hypersensitivity or prior reaction to any of the formulation excipients in the study drugs.
13. History of stage III or greater cancer, excluding urothelial cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of registration. Subjects with a history of stage I or II cancer, must have been adequately treated and have been disease-free for ≥ 3 years at the time of registration.
14. Concomitant active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis)
15. Progressive viral or bacterial infection
16. All infections must be resolved and the patient must remain afebrile for seven days without antibiotics prior to being placed on study
17. Any underlying medical condition that, in the Investigator's opinion, will make the administration of study vaccine hazardous to the patient, would obscure the interpretation of adverse events, or not permit adequate surgical resection.
18. Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Complete Response Proportion (CR) | 9 months (Phase II)
  'CR' Proportion is confirmed by negative biopsy, cystoscopy, cytology weekly times 2 with the first assessment three months after first intravesical treatment and then assessed again at 9 month. Two consecutive positive urine cytologies to confirm a persistent or recurrent disease if visual and biopsy is negative. Random biopsy mandatory at the first assessment in the trigone, bladder dome, right, left , anterior and posterior of the bladder wall.
Durable Complete Response Proportion (DCR) | 15 months (Phase III)
  DCR proportion of DCR lasting 12 months or longer will be conducted after a follow up period of 15 months for each patient. The first complete response assessment will be at 3 month.

SECONDARY OUTCOMES:
Progression rate to muscle invasive disease | Throughout the study with expected average of 12 months
  The Progression rate to muscle invasive disease rate is based on analysis from comparing disease status at the time of enrollment versus disease status (for those patients with muscle invasion) at the time of cystectomy or TURBT
Complete Response Survival | 15 months
  The Complete Response Survival time to events of patients who have achieved a complete response at the 3 month assessment will be compared with a log rank test.
Safety Events | Expected average of two years throughout the study
  The number and percentage of patients experiencing one or more adverse events will be summarized by relationship to study drug, and severity.
Cystectomy Free Survival | 15 month
  The Cystectomy Free Survival time to events of patients will be compared with a log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Alex W Yeung, MBBS, Study Chair — CG Oncology, Inc.
Locations (7):
- United States (7):
  - BCG Oncology, Phoenix, Arizona
  - University of California, San Diego- Moores Cancer Center, La Jolla, California
  - UCLA Institute of Urological Oncology, Los Angeles, California
  - University of California, Davis- Cancer Center, Sacramento, California
  - University of Chicago, Department of Surgery, Section of Urology, Chicago, Illinois
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center Department of Urologic Surgery, Nashville, Tennessee